CLINICAL TRIAL: NCT04885335
Title: Evaluation of the Management of Acute Appendicitis Before Emergency Department in Children: a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: BAlouhhey_appendicites
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PAS (Pediatric Appendicitis Score) survey — Score ≤ 5: appendicitis unlikely. Score ≥ 6: probable appendicitis. core ≥ 7: very probable appendicitis

SUMMARY:
Acute appendicitis is the first visceral surgical emergency in pediatrics with about 30,000 cases in children having been described in France.

It concerns 0.3% of children under 15 with a maximum frequency between 8 and 13 years of age. Acute appendicitis has a significant morbidity rate of 8% and a mortality rate under 0.1%.

10 to 25% of the children admitted to emergency rooms for abdominal pain have appendicitis.

In 20 to 30% of the cases, the initial symptoms are atypical, which explains the difficulty in diagnosing.

The purpose of our study is to evaluate the quality of general practitioners in the diagnosis of acute appendicitis, its severity and the diagnostic criteria used.

Furthermore, it is not as easy to evaluate pain or examine a complaint in children as it is in adults.

Appendicectomy is the treatment of choice for all acute appendicitis. The importance of early diagnosis and treatment is, therefore, essential. Many predictive diagnostic scores have been studied over the years. The Pediatric Appendicitis Score (PAS) using typical symptoms of acute appendicitis and biological items was published in 2002. Nowadays, it is still considered as a reference and has been validated by other studies.

Most of the patients suffering from abdominal pain first consult their general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Child <16 years
* abdominal symptoms
* consulting in the pediatric emergency department of Limoges University center.

Exclusion Criteria:

* Child >=16 years

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: -Child <16 years with abdominal symptoms and consulting in the pediatric emergency department of Limoges University center.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
PAS score | At 5 month
  Score ≤ 5: appendicitis unlikely. Score ≥ 6: probable appendicitis. Score ≥ 7: very probable appendicitis

SECONDARY OUTCOMES:
Surgery for appendicitis | At 5 month

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric emergency department, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vevaud K, Dallocchio A, Dumoitier N, Laspougeas A, Labrunie A, Belgacem A, Fourcade L, Ballouhey Q. A prospective study to evaluate the contribution of the pediatric appendicitis score in the decision process. BMC Pediatr. 2024 Feb 19;24(1):131. doi: 10.1186/s12887-024-04619-z. PMID 38373918